CLINICAL TRIAL: NCT03231813
Title: Regional Differences of Cutaneous Irritation and Its Effect on Skin Barrier Recovery: A Randomised, Controlled Trial
Brief Title: Regional Differences of Cutaneous Irritation and Its Effect on Skin Barrier Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 003-08/17-03/0001
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-06

CONDITIONS: Irritant Contact Dermatitis
Keywords: irritant contact dermatitis; sodium lauryl sulphate; emollients; transepidermal water loss
MeSH Terms: conditions — Dermatitis, Irritant | interventions — Emollients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SLS irritation model and Treatment (Experimental): SLS induced irritation on two sites each on forearms and back Emollient cream treatment
  Interventions: Procedure: Sodium lauryl sulphate induced irritation; Other: Emollient, moisturizing cream
- SLS irritation model and No Treatment (Placebo Comparator): SLS induced irritation on two sites each on forearms and back No treatment
  Interventions: Procedure: Sodium lauryl sulphate induced irritation
- Sham irritation and Treatment (Sham Comparator): Sham irritation (water) on two sites each on forearms and back Emollient cream treatment
  Interventions: Other: Emollient, moisturizing cream
- Sham irritation and No Treatment (No Intervention): Sham irritation (water) on two sites each on forearms and back No treatment

INTERVENTIONS:
Procedure: Sodium lauryl sulphate induced irritation — Sodium lauryl sulphate will be applied to specified skin sites according to randomization protocol to induce irritation. 60 uL of 2% w/v SLS will be applied to skin under occlusion by large Finn chamber for 24 hours as described in the guidelines by Standardization group of European Society of Contact Dermatitis.
  Arms: SLS irritation model and No Treatment; SLS irritation model and Treatment
Other: Emollient, moisturizing cream — Commercially available topical emollient cream will be applied by each participant to treatment sites according to randomization protocol.
  Arms: SLS irritation model and Treatment; Sham irritation and Treatment

SUMMARY:
Irritant contact dermatitis induced by sodium lauryl sulphate (SLS) is often used as a model for testing efficacy of various topical preparations. Aforementioned model is standardized and described in guidelines, but it is not explicitly stated where the irritation should be induced. Published clinical trials usually irritate volar aspect of forearms or upper back. Also, lower back and dorsal aspect of forearm are sometimes used.

Skin parameters vary depending on anatomic location of measured skin. There is a difference in stratum corneum thickness, hydration and transepidermal water loss across different locations, including between volar forearm and upper back.

Furthermore, regional difference in skin response to irritation by tape stripping and benzalkonium chloride were observed. Such differences are also possible in SLS irritation model. One study has shown higher, but not statistically significant, response of back in comparison to forearms, but it had a very small sample size (n=9).

Moreover, there are regional variations of topical preparations absorption. Hydrocortisone had 1,7 times higher absorption when applied to upper back in comparison to forearms. Those variations could be explained by different corneocyte size and number of their layers between back and hands.

Skin baseline properties and response to irritation seem to be dependent on anatomic position. Those differences could mean different response to treatment. Since published trials only tested efficacy of various preparations on one anatomic location, it is possible their results would be different if tested on other body parts. It could limit validity and usefulness of conducted trials. The aim of this study is to determine if there are regional differences of skin response to irritation and emollient cream treatment in irritant contact dermatitis model.

ELIGIBILITY:
Inclusion Criteria:

* young, healthy volunteers who gave written informed consent

Exclusion Criteria:

* skin disease, skin damage on measurement sites, use of corticosteroids and immunomodulators a month prior the inclusion and during the trial, use of emollients three days prior the inclusion in the trial, non-adherence to the trial protocol, exposure to artificial UV radiation, pregnancy and lactation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss | Five measurements; baseline, irritation, first, third and ninth day of treatment
  Tewameter will be used to assess skin barrier function as a measurement of the water loss (g/hm2).
Stratum corneum hydration | Five measurements; baseline, irritation, first, third and ninth day of treatment
  Corneometer will be used to estimate skin dryness. It is a relative measurement and uses arbitrary units (AU).
Erythema | Five measurements; baseline, irritation, first, third and ninth day of treatment
  Mexameter will be used to assess erythema. It is a relative measurement and uses arbitrary units (AU).

SECONDARY OUTCOMES:
Clinical score | Five assessments: baseline, irritation, first, third and ninth day of treatment
  Skin response to irritation and treatment will be assessed using a five-point scale to describe changes in skin erythema, roughness, scaling, oedema, and fissures.

CONTACTS AND LOCATIONS:
Overall Officials: Dario Leskur, MPharm, Principal Investigator — University of Split, School of Medicine
Locations (1):
- School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tupker RA, Willis C, Berardesca E, Lee CH, Fartasch M, Agner T, Serup J. Guidelines on sodium lauryl sulfate (SLS) exposure tests. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1997 Aug;37(2):53-69. doi: 10.1111/j.1600-0536.1997.tb00041.x. PMID 9285167
- [Background] Wilhelm KP, Cua AB, Maibach HI. Skin aging. Effect on transepidermal water loss, stratum corneum hydration, skin surface pH, and casual sebum content. Arch Dermatol. 1991 Dec;127(12):1806-9. doi: 10.1001/archderm.127.12.1806. PMID 1845280
- [Background] Schwindt DA, Wilhelm KP, Maibach HI. Water diffusion characteristics of human stratum corneum at different anatomical sites in vivo. J Invest Dermatol. 1998 Sep;111(3):385-9. doi: 10.1046/j.1523-1747.1998.00321.x. PMID 9740228
- [Background] Lee CH, Maibach HI. The sodium lauryl sulfate model: an overview. Contact Dermatitis. 1995 Jul;33(1):1-7. doi: 10.1111/j.1600-0536.1995.tb00438.x. PMID 7493454
- [Background] Tagami H. Location-related differences in structure and function of the stratum corneum with special emphasis on those of the facial skin. Int J Cosmet Sci. 2008 Dec;30(6):413-34. doi: 10.1111/j.1468-2494.2008.00459.x. PMID 19099543
- [Background] Nedelec B, Forget NJ, Hurtubise T, Cimino S, de Muszka F, Legault A, Liu WL, de Oliveira A, Calva V, Correa JA. Skin characteristics: normative data for elasticity, erythema, melanin, and thickness at 16 different anatomical locations. Skin Res Technol. 2016 Aug;22(3):263-75. doi: 10.1111/srt.12256. Epub 2015 Sep 1. PMID 26333046
- [Background] Darlenski R, Fluhr JW. Influence of skin type, race, sex, and anatomic location on epidermal barrier function. Clin Dermatol. 2012 May-Jun;30(3):269-73. doi: 10.1016/j.clindermatol.2011.08.013. PMID 22507039
- [Background] Berardesca E, Distante F. The modulation of skin irritation. Contact Dermatitis. 1994 Nov;31(5):281-7. doi: 10.1111/j.1600-0536.1994.tb02019.x. PMID 7867323
- [Background] Emtestam L, Ollmar S. Electrical impedance index in human skin: measurements after occlusion, in 5 anatomical regions and in mild irritant contact dermatitis. Contact Dermatitis. 1993 Feb;28(2):104-8. doi: 10.1111/j.1600-0536.1993.tb03352.x. PMID 8458202
- [Background] Cua AB, Wilhelm KP, Maibach HI. Frictional properties of human skin: relation to age, sex and anatomical region, stratum corneum hydration and transepidermal water loss. Br J Dermatol. 1990 Oct;123(4):473-9. doi: 10.1111/j.1365-2133.1990.tb01452.x. PMID 2095179
- [Background] Kleesz P, Darlenski R, Fluhr JW. Full-body skin mapping for six biophysical parameters: baseline values at 16 anatomical sites in 125 human subjects. Skin Pharmacol Physiol. 2012;25(1):25-33. doi: 10.1159/000330721. Epub 2011 Sep 7. PMID 21912200
- [Background] Lavrijsen AP, Geelen FA, Oestmann E, Hermans J, Bodda HE, Ponec M. Comparison of human back versus arm skin region for its suitability to test weak irritants. Skin Res Technol. 1996 May;2(2):70-7. doi: 10.1111/j.1600-0846.1996.tb00062.x. PMID 27327221
- [Background] Holbrook KA, Odland GF. Regional differences in the thickness (cell layers) of the human stratum corneum: an ultrastructural analysis. J Invest Dermatol. 1974 Apr;62(4):415-22. doi: 10.1111/1523-1747.ep12701670. No abstract available. PMID 4820685
- [Background] Hadgraft J, Lane ME. Transepidermal water loss and skin site: a hypothesis. Int J Pharm. 2009 May 21;373(1-2):1-3. doi: 10.1016/j.ijpharm.2009.02.007. Epub 2009 Feb 21. PMID 19429281
- [Background] Ya-Xian Z, Suetake T, Tagami H. Number of cell layers of the stratum corneum in normal skin - relationship to the anatomical location on the body, age, sex and physical parameters. Arch Dermatol Res. 1999 Oct;291(10):555-9. doi: 10.1007/s004030050453. PMID 10552214
- [Background] Fluhr JW, Dickel H, Kuss O, Weyher I, Diepgen TL, Berardesca E. Impact of anatomical location on barrier recovery, surface pH and stratum corneum hydration after acute barrier disruption. Br J Dermatol. 2002 May;146(5):770-6. doi: 10.1046/j.1365-2133.2002.04695.x. PMID 12000372
- [Background] Breternitz M, Flach M, Prassler J, Elsner P, Fluhr JW. Acute barrier disruption by adhesive tapes is influenced by pressure, time and anatomical location: integrity and cohesion assessed by sequential tape stripping. A randomized, controlled study. Br J Dermatol. 2007 Feb;156(2):231-40. doi: 10.1111/j.1365-2133.2006.07632.x. PMID 17223861
- [Background] Magnusson B, Hersle K. Patch test methods. II. Regional variations of patch test responses. Acta Derm Venereol. 1965;45(4):257-61. No abstract available. PMID 4162958
- [Background] Cua AB, Wilhelm KP, Maibach HI. Cutaneous sodium lauryl sulphate irritation potential: age and regional variability. Br J Dermatol. 1990 Nov;123(5):607-13. doi: 10.1111/j.1365-2133.1990.tb01477.x. PMID 2248890
- [Background] Feldmann RJ, Maibach HI. Regional variation in percutaneous penetration of 14C cortisol in man. J Invest Dermatol. 1967 Feb;48(2):181-3. doi: 10.1038/jid.1967.29. No abstract available. PMID 6020682
- [Background] Rougier A, Dupuis D, Lotte C, Roguet R, Wester RC, Maibach HI. Regional variation in percutaneous absorption in man: measurement by the stripping method. Arch Dermatol Res. 1986;278(6):465-9. doi: 10.1007/BF00455165. PMID 3789805
- [Background] Rougier A, Lotte C, Maibach HI. In vivo percutaneous penetration of some organic compounds related to anatomic site in humans: predictive assessment by the stripping method. J Pharm Sci. 1987 Jun;76(6):451-4. doi: 10.1002/jps.2600760608. PMID 3625489
- [Background] Machado M, Salgado TM, Hadgraft J, Lane ME. The relationship between transepidermal water loss and skin permeability. Int J Pharm. 2010 Jan 15;384(1-2):73-7. doi: 10.1016/j.ijpharm.2009.09.044. Epub 2009 Sep 30. PMID 19799976
- [Derived] Leskur D, Bukic J, Petric A, Zekan L, Rusic D, Seselja Perisin A, Petric I, Stipic M, Puizina-Ivic N, Modun D. Anatomical site differences of sodium lauryl sulfate-induced irritation: randomized controlled trial. Br J Dermatol. 2019 Jul;181(1):175-185. doi: 10.1111/bjd.17633. Epub 2019 Apr 11. PMID 30637727